CLINICAL TRIAL: NCT04126941
Title: Bi-daily Injection of Subcutaneous Teriparatide in Children With Hypoparathyroidism: Single-center Experience
Brief Title: Monocentric Study on the Use of Teriparatide in Children With hypoparathyroïdism
Acronym: FOR-HYPO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2019 FOR-HYPO
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Hypoparathyroidism
Keywords: Hypoparathyroidism; Teriparatide
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Teriparatide: Patients with hypoparathyroidism treated by teriparatide
  Interventions: Other: Serum calcium concentrations results

INTERVENTIONS:
Other: Serum calcium concentrations results — To compare serum calcium concentrations results in patients with hypoparathyroidism before and three months after initiation of teriparatide therapy

SUMMARY:
Pediatric hypoparathyroidism is an orphan disease. Conventional management combines native and active vitamin D, calcium supplementation and sometimes phosphate binders, with the risk of long term hypercalciuria, nephrocalcinosis and further renal impairment. The use of teriparatide has been reported in adults (daily or bi-daily subcutaneous infusions) and in children (rather continuous subcutaneous infusion) as second-line therapy.

The objective of this study is to obtain efficacy and safety data on the use of teriparatide in children with hypoparathyroidism to improve our knowledge of their management.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypoparathyroidism
* Patients treated with teriparatide
* Patients followed in the reference center for calcium and phosphate metabolism diseases of Lyon.
* For children under 18: patient and parent (s) / parent having been informed of the study and having expressed their non-opposition

Exclusion Criteria:

* No social security support

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with hypoPTH (Hypoparathyroidism) treated with teriparatide
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Serum calcium concentration | 3 months after treatment initiation

SECONDARY OUTCOMES:
Serum calcium concentration | 1 month after treatment initiation
Serum calcium concentration | 6 months after treatment initiation
Serum calcium concentration | 12 months after treatment initiation
Serum calcium concentration | 3 years after treatment initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Néphrologie, Rhumatologie et Dermatologie Pédiatriques - Hôpital Femme Mère Enfant, Bron, France